CLINICAL TRIAL: NCT00382460
Title: Pravastatin or Atorvastatin Evaluation and Infection Therapy (TIMI22)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: CV123-229; TIMI22
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Actue Coronary Syndromes
MeSH Terms: interventions — Pravastatin

INTERVENTIONS:
Drug: PRAVASTATIN SODIUM

SUMMARY:
The primary purpose of the study was to evaluate 4000 subjects with acute coronary syndrome by comparing pravastatin 40 mg to atorvastatin 80 mg to determine if they are clinically equivalent, and to evaluate the effectiveness of gatifloxacin therapy in reducing cardiovascular events in combination with statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for MI or high risk unstable angina within the last 10 days.
* Total cholesterol 240 mg/dl or greater.
* Stabilized post ACS

Exclusion Criteria:

* Co-morbidity with life expectations no more than 2 years.
* Current lipid lowering therapy
* Corrected QT interval
* Need for Class IA or III antiarrhythmic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2000-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate the clinical equivalence of pravastatin 40 mg and atorvastatin 80 mg in reducing death or major cardiovascular event after 2 years
To demonstrate in subjects with ACS that Gatifloxacin is effective in reducing death or major cardiovascular event after 2 years, compared to placebo.

SECONDARY OUTCOMES:
To compare the risk of nonfatal MI or coronary heart disease death between pravastatin and atorvastatin, and gatifloxacin and placebo.

REFERENCES:
- [Derived] Mengozzi A, Trico D, Natali A. A novel method for interpreting survival analysis data: description and test on three major clinical trials on cardiovascular prevention. Trials. 2020 Jun 26;21(1):578. doi: 10.1186/s13063-020-04511-y. PMID 32586346
- [Derived] Bonaca MP, O'Malley RG, Jarolim P, Scirica BM, Murphy SA, Conrad MJ, Cannon CP, White HD, Braunwald E, Morrow DA, Sabatine MS. Serial Cardiac Troponin Measured Using a High-Sensitivity Assay in Stable Patients With Ischemic Heart Disease. J Am Coll Cardiol. 2016 Jul 19;68(3):322-323. doi: 10.1016/j.jacc.2016.04.046. No abstract available. PMID 27417011
- [Derived] Nazer B, Ray KK, Murphy SA, Gibson CM, Cannon CP. Urinary albumin concentration and long-term cardiovascular risk in acute coronary syndrome patients: a PROVE IT-TIMI 22 substudy. J Thromb Thrombolysis. 2013 Oct;36(3):233-9. doi: 10.1007/s11239-012-0853-0. PMID 23212806
- [Derived] Wilson SR, Sabatine MS, Wiviott SD, Ray KK, De Lemos JA, Zhou S, Rifai N, Cannon CP, Morrow DA; TIMI Study Group. Assessment of adiponectin and the risk of recurrent cardiovascular events in patients presenting with an acute coronary syndrome: observations from the Pravastatin Or atorVastatin Evaluation and Infection Trial-Thrombolysis in Myocardial Infarction 22 (PROVE IT-TIMI 22). Am Heart J. 2011 Jun;161(6):1147-55.e1. doi: 10.1016/j.ahj.2011.02.014. Epub 2011 May 11. PMID 21641362
- [Derived] Truong QA, Murphy SA, McCabe CH, Armani A, Cannon CP; TIMI Study Group. Benefit of intensive statin therapy in women: results from PROVE IT-TIMI 22. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):328-36. doi: 10.1161/CIRCOUTCOMES.110.957720. Epub 2011 Apr 12. PMID 21487089
- [Derived] Nazer B, Ray KK, Sloan S, Scirica B, Morrow DA, Cannon CP, Braunwald E. Prognostic utility of neopterin and risk of heart failure hospitalization after an acute coronary syndrome. Eur Heart J. 2011 Jun;32(11):1390-7. doi: 10.1093/eurheartj/ehr032. Epub 2011 Feb 22. PMID 21345849
- [Derived] Bangalore S, Qin J, Sloan S, Murphy SA, Cannon CP; PROVE IT-TIMI 22 Trial Investigators. What is the optimal blood pressure in patients after acute coronary syndromes?: Relationship of blood pressure and cardiovascular events in the PRavastatin OR atorVastatin Evaluation and Infection Therapy-Thrombolysis In Myocardial Infarction (PROVE IT-TIMI) 22 trial. Circulation. 2010 Nov 23;122(21):2142-51. doi: 10.1161/CIRCULATIONAHA.109.905687. Epub 2010 Nov 8. PMID 21060068
- [Derived] Gibson CM, Pride YB, Hochberg CP, Sloan S, Sabatine MS, Cannon CP; TIMI Study Group. Effect of intensive statin therapy on clinical outcomes among patients undergoing percutaneous coronary intervention for acute coronary syndrome. PCI-PROVE IT: A PROVE IT-TIMI 22 (Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis In Myocardial Infarction 22) Substudy. J Am Coll Cardiol. 2009 Dec 8;54(24):2290-5. doi: 10.1016/j.jacc.2009.09.010. PMID 19958964
- [Derived] Giraldez RR, Giugliano RP, Mohanavelu S, Murphy SA, McCabe CH, Cannon CP, Braunwald E. Baseline low-density lipoprotein cholesterol is an important predictor of the benefit of intensive lipid-lowering therapy: a PROVE IT-TIMI 22 (Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis In Myocardial Infarction 22) analysis. J Am Coll Cardiol. 2008 Sep 9;52(11):914-20. doi: 10.1016/j.jacc.2008.05.046. PMID 18772061
- [Derived] Miller M, Cannon CP, Murphy SA, Qin J, Ray KK, Braunwald E; PROVE IT-TIMI 22 Investigators. Impact of triglyceride levels beyond low-density lipoprotein cholesterol after acute coronary syndrome in the PROVE IT-TIMI 22 trial. J Am Coll Cardiol. 2008 Feb 19;51(7):724-30. doi: 10.1016/j.jacc.2007.10.038. PMID 18279736